CLINICAL TRIAL: NCT02277418
Title: Intubation of Child and Infant Manikins During Resuscitation. Does the Venner™ A.P. Advance™ Video Laryngoscope Improve Nurses' Performance?
Brief Title: Venner a.p. Advance Video Laryngoscope
Acronym: VAVL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/05
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Intubation; Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Child ETI withoutchest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation without chest compressions.
  Interventions: Device: VAVL; Device: MIL
- Child ETI with chest compressions (Experimental): Endotracheal intubation of mannikin during resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: VAVL; Device: MIL
- Infant ETI with chest compressions (Experimental): endotracheal intubation (ETI) during infant mannikin resuscitation with uninterrupted chest compressions.
  Interventions: Device: VAVL; Device: MIL
- Infant ETI without chest compressions (Experimental): Endotracheal intubation of infant mannikin during resuscitation without chest compressions.
  Interventions: Device: VAVL; Device: MIL

INTERVENTIONS:
Device: VAVL — Videolaryngoscope
  Other Names: Venner a.p. advance video laryngoscope
Device: MIL — Direct laryngoscopy
  Other Names: Miller Laryngoscope

SUMMARY:
The purpose of this study was to compare the Venner a.p. advance video laryngoscope to Miller laryngoscope during resuscitation with and without chest compressions.

DETAILED DESCRIPTION:
Endotracheal intubation (ETI) is a life-saving procedure performed daily in emergency medicine. The European Resuscitation Council (ERC) 2010 cardiopulmonary resuscitation (CPR) guidelines suggest that intubators should be able to secure the airway without interrupting chest compression. However, ETI with uninterrupted chest compression in patients can be a very difficult skill to acquire.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel (paramedics, nurses, physicians

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Time to intubation | 1 day
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.

SECONDARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.
POGO score | 1 day
  self-reported percentage of glottis opening (POGO) score
VAS score | 1 day
  participants were asked which method they would prefer in a real-life resuscitation.
Cormack-Lehan scale | 1 day
  self reported Cormack-Lehan scale during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland